CLINICAL TRIAL: NCT03878719
Title: A Multicenter, Open-label Phase 1b Study of the Combination of Binimetinib and Encorafenib in Adolescent Patients With Unresectable or Metastatic BRAF V600-mutant Melanoma
Brief Title: Study of the Combination of Binimetinib and Encorafenib in Adolescent Patients With Unresectable or Metastatic BRAF V600-mutant Melanoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: The trial was terminated early on 05 October 2022 due to non-feasibility and poor recruitment and not based on safety concerns.
Sponsor: Pfizer (Industry)
Collaborators: Pierre Fabre Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARRAY-162-115; C4221011 (Other: Alias Study Number); 2018-001946-32 (EudraCT Number)
Record Dates: First submitted 2019-02-20; First posted 2019-03-18 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Melanoma
Keywords: Adolescent; BRAF V600K; BRAF V600E
MeSH Terms: conditions — Melanoma | interventions — binimetinib; encorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Safety Run-in Phase (Experimental): * binimetinib taken twice daily (BID) and
  * encorafenib taken once daily (QD)
  Dose levels by patient body surface area (BSA) for binimetinib and encorafenib tablets/capsules are specified in the protocol.
  Interventions: Drug: binimetinib; Drug: encorafenib
- Expansion Phase (Experimental): * binimetinib taken twice daily (BID) and
  * encorafenib taken once daily (QD)
  Dose levels by patient body surface area (BSA) for binimetinib and encorafenib tablets/capsules and pediatric formulations are specified in the protocol.
  Interventions: Drug: binimetinib; Drug: encorafenib

INTERVENTIONS:
Drug: binimetinib — taken orally
Drug: encorafenib — taken orally

SUMMARY:
This is a multicenter Phase 1b, open-label study to evaluate the pharmacokinetic, safety and efficacy of binimetinib and encorafenib co-administered to adolescent patients with BRAF V600-mutant advanced/metastatic melanoma. The study consists of a Safety Run-in Phase to determine the RDE (recommended dose in expansion), followed by an Expansion Phase.

DETAILED DESCRIPTION:
The study did not recruit the desired number of subjects and as a result does not have sufficient data for quantitative statistical analyses. Additionally, results data cannot be reported because doing so would risk re-identification of the participant.

ELIGIBILITY:
Key Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for enrollment in the study.

* Histologically confirmed diagnosis of locally advanced, unresectable or metastatic cutaneous melanoma or unknown primary melanoma American Joint Committee on Cancer Stage IIIB, IIIC, or IV.
* Presence of BRAF V600E or V600K mutation in tumor tissue as determined by a local or central laboratory
* Adequate cardiac function:

  * Left ventricular ejection fraction (LVEF) ≥ 50% as determined by ECHO or multi-gated acquisition (MUGA) scan and above the institutional lower limit of normal (LLN);
  * Triplicate average baseline QTcF value ≤ 450 ms.
* Adequate bone marrow, organ function, and laboratory parameters:

  * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L;
  * Hemoglobin ≥ 9 g/dL with or without transfusions;
  * Platelets ≥ 75 × 10⁹/L without transfusions;
  * Aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) ≤ 2.5 × upper limit of normal (ULN); in patients with liver metastases ≤ 5 × ULN;
  * Total bilirubin ≤ 1.5 × ULN;
  * Creatinine ≤ 1.5 × institutional ULN for age, or calculated creatinine clearance ≥ 70 mL/min/1.73 m² (following Schwartz formula).
* Adequate performance status at Screening:

  * Patients < 16 years old: Lansky Performance Scale score ≥ 80
  * Patients 16 to 17 years old: Karnofsky Performance Scale score ≥ 80

Key Exclusion Criteria:

Patients meeting any of the following criteria are not eligible for enrollment in the study.

* Uveal or mucosal melanoma.
* Brain metastases that are uncontrolled or symptomatic, require steroids, are potentially life-threatening or have required radiation within 28 days prior to starting study drug.
* History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO
* Prior therapy with a BRAF inhibitor (e.g., dabrafenib, vemurafenib) and/or a MEK inhibitor (e.g., trametinib, cobimetinib).
* Impaired cardiovascular function or clinically significant cardiovascular disease, including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) < 6 months prior to screening,
  * Symptomatic chronic heart failure, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality < 6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia.
* Concurrent neuromuscular disorder associated with elevated creatine kinase (CK)
* Uncontrolled arterial hypertension despite medical treatment
* Presence of BRAFʷͭ or indeterminate melanoma in tumor tissue.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1 (Actual)
Dates: Start 2020-08-03 (Actual); Primary Completion 2022-08-19 (Actual); Study Completion 2022-08-19 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) parameter (time to reach the maximum observed plasma concentration Cmax [Tmax]) for binimetinib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Cmax) for binimetinib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (time of last PK sample [Tlast]) for binimetinib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (area under the plasma concentration-time curve from time zero to Tlast [AUClast]) for binimetinib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tmax) for binimetinib's active metabolite (AR00426032) | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Cmax) for AR00426032 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tlast) for AR00426032 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (AUClast) for AR00426032 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tmax) for encorafenib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Cmax) for encorafenib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tlast) for encorafenib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (AUClast) for encorafenib | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tmax) for encorafenib's metabolite (LHY746) | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Cmax) for LHY746 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (Tlast) for LHY746 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (AUClast) for LHY746 | Day 1 and Day 15 of Cycle 1, 28 day cycles
PK parameter (trough concentration [Ctrough]) for binimetinib | at time zero Day 15 of Cycle 1, 28 day cycles
PK parameter (trough concentration [Ctrough]) for binimetinib | at time zero Day 1 of Cycle 2, 28 day cycles
PK parameter (trough concentration [Ctrough]) for binimetinib | at time zero Day 1 of Cycle 3, 28 day cycles
PK parameter (Ctrough) for AR00426032 | at time zero Day 15 of Cycle 1, 28 day cycles
PK parameter (Ctrough) for AR00426032 | at time zero Day 1 of Cycle 2, 28 day cycles
PK parameter (Ctrough) for AR00426032 | at time zero Day 1 of Cycle 3, 28 day cycles
PK parameter (Ctrough) for encorafenib | at time zero Day 15 of Cycle 1, 28 day cycles
PK parameter (Ctrough) for encorafenib | at time zero Day 1 of Cycle 2, 28 day cycles
PK parameter (Ctrough) for encorafenib | at time zero Day 1 of Cycle 3, 28 day cycles
PK parameter (Ctrough) for LHY746 | at time zero Day 15 of Cycle 1, 28 day cycles
PK parameter (Ctrough) for LHY746 | at time zero Day 1 of Cycle 2, 28 day cycles
PK parameter (Ctrough) for LHY746 | at time zero Day 1 of Cycle 3, 28 day cycles

SECONDARY OUTCOMES:
Incidence and severity of adverse events (AEs) | From informed consent up to 30 days following last dose of study drug
Incidence of dose-limiting toxicities (DLTs) | Duration of treatment for safety run-in phase, approximately 6 months, 28 day cycles
Palatability score for the pediatric formulations as assessed by an age-appropriate questionnaire for binimetinib | Through Cycle 3 Day 1 in patients receiving the pediatric formulations in the Expansion Phase, 28 day cycles
  Five-point Hedonic scale from 1 to 5, 5=really good
Palatability score for the pediatric formulations as assessed by an age-appropriate questionnaire for encorafenib | Through Cycle 3 Day 1 in patients receiving the pediatric formulations in the Expansion Phase, 28 day cycles
  Five-point Hedonic scale from 1 to 5, 5=really good
Objective response rate (ORR) assessed by the investigator, based on Response Criteria Evaluation in Solid Tumors (RECIST) v1.1 | Duration of treatment, approximately 6 months, 28 day cycles
Duration of response (DOR) | Duration of treatment, approximately 6 months, 28 day cycles
Time to response | Duration of treatment, approximately 6 months, 28 day cycles
Progression-free survival (PFS) | Duration of treatment, approximately 6 months, 28 day cycles
One-year survival rate | From first dose up to 1 year after treatment initiation
Change from baseline bone age and the difference in bone age and chronological age | Duration of treatment, approximately 6 months, 28 day cycles
Change from Baseline in bone densitometry based on dual energy X-ray absorptiometry (DEXA) scan. | Duration of treatment, approximately 6 months, 28 day cycles
Change from Baseline in calcium-phosphorus product (Ca × P) | Duration of treatment, approximately 6 months, 28 day cycles

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Fondazione IRCCS Istituto Nazionale Dei Tumori, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=ARRAY-162-115